CLINICAL TRIAL: NCT05441020
Title: Development, Feasibility Testing and Validation of a Survey Set to Measure Patient-Reported Outcomes Among Hemodialysis Patients in Turkey
Acronym: DOPRO
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: acromion GmbH (Industry); Vector Psychometric Group, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: HD-HOME-01-TR
Record Dates: First submitted 2022-05-18; First posted 2022-07-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Hemodialysis; Psychometric tests; Patient questionnaire
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Administration of patient questionnaire — Patients undergoing maintenance hemodialysis complete electronic questionnaires on a tablet computer during this study to assess patient reported outcomes.

SUMMARY:
Development, feasibility testing and validation of a Survey Set to Measure Patient-Reported Outcomes among Hemodialysis Patients in Turkey: Creating and testing an electronic patient questionnaire that is suitable to measure health-related quality of life in Turkish dialysis patients in clinical as well as in home care settings.

DETAILED DESCRIPTION:
Individuals with chronic kidney disease represent a growing population in adult and pediatric practices. This has resulted in a drive to optimize patient care and outcomes. Historically, healthcare outcomes focused on morbidity, mortality or complication rates, but failed to provide meaningful data on the value of medicine to patients and the quality of life gained or lost. Several studies have revealed that treatments aimed at minimizing morbidity and mortality in end-stage renal disease (ESRD) have very often been ineffective. Therefore, attention to HRQOL among ESRD patients is crucial.

The aim of this pilot study is creating and testing an electronic patient questionnaire that is suitable to measure health-related quality of life in Turkish dialysis patients. This questionnaire consists of the PROMIS Cognitive Function and Abilities Subset, the PROMIS-29, a new post-dialysis recovery time module, the MOS-Social Support Scale (MOS-SSS), Subscales of the KDQOL SF 1.3 (sexual function & cognitive function), the General Self-Efficacy Scale and the Health Services Utilization And Productivity Loss Survey which are to be delivered together on a tablet computer.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorized physician
* Age of 18 -80 years
* Ability to understand the nature and requirements of the study
* Literacy in Turkish including the ability to read with regards to visual acuity and the ability to understand what is read
* General ability to use a tablet (the study nurse will instruct the patient how to use the study-tablet during the conduct of the study)
* To be on stable maintenance hemodialysis (HD) for over 3 months (prevalent patients)

Exclusion Criteria:

* Any conditions which could interfere with the patient's ability to comply with the study
* Previous participation in the same study
* Participation in an interventional clinical study during the preceding 30 days
* Serious life-limiting co-morbid situations, namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease, which causes life-expectancy less than a year,
* Acute cardiovascular events including myocardial infarction, stroke and unstable angina pectoris requiring hospitalization within the last 6 months,
* To have cognitive or mental co-morbidities which prevent reliable answering of questions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish dialysis patients (in center or home dialysis)
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Validation of Patient Reported Outcome Measures Information System-29 (PROMIS-29) | 2 weeks between test and retest
Translating and testing PROMIS Cognitive Function and Abilities Subscale (PROMIS-CFS) | 2 weeks between test and retest
Translating and testing feasibility of a new post-dialysis recovery time module adapted from PROMIS scale on fatigue | Single Administration in cross-sectional design
Testing feasibility and usefulness of measuring Social Support, potential reduction of items and internal consistency of the MOS-Social Support Scale (MOS-SSS) | Single Administration in cross-sectional design
Assessing feasibility and usefulness of measuring General Self-Efficacy Scale (GSE) | Single Administration in cross-sectional design
Testing feasibility of the Telephone Cognitive Screen (T-Cog-S) | Single Administration in cross-sectional design
Testing feasibility of the kidney disease targeted subscales (sexual function & cognitive function) of the Kidney Disease Quality of Life Short Form Version 1.3 (KDQOL SF 1.3) | Single Administration in cross-sectional design
Testing feasibility of Health Services Utilization and Productivity Loss Survey | Single Administration in cross-sectional design

CONTACTS AND LOCATIONS:
Overall Officials: Hayriye Elbi, Prof Dr, Principal Investigator — Ege University Medical Faculty
Locations (7):
- Turkey (Türkiye) (7):
  - Fresenius Nefroloji Hizmetleri A.Ş.-Bornova Branch, Izmir
  - Fresenius Nefroloji Hizmetleri A.Ş.-Buca Branch, Izmir
  - Fresenius Nefroloji Hizmetleri A.Ş.-İzmir Üçkuyular Branch, Izmir
  - Fresenius Nefroloji Hizmetleri A.Ş.-İzmir Hatay Branch, Izmir
  - İzmir Renal Özel Sağlık Tesisleri ve Malzemeleri Sanayi Tic. A.Ş- Yeşilyurt Branch, Izmir
  - Gaziemir Özel Sağlık Hizmetleri Tesisleri Malzemeleri Sanayi ve Tic. A.Ş. - Gaziemir Branch, Izmir
  - Fresenius Nefroloji Hizmetleri A.Ş.-Karşıyaka Branch, Izmir